CLINICAL TRIAL: NCT05474859
Title: A Phase 1, Multicenter Tolerability and Pharmacokinetic Study of Ascending Continuous Oral Doses of XT-0528 in Subjects With Advanced or Metastatic Solid Tumor Malignancies
Brief Title: Subjects With Advanced or Metastatic Solid Tumor Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xenthera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XT-001
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Solid Tumor; Advanced Solid Tumor
Keywords: Interleukin 17 (IL17); retinoic acid related orphan nuclear receptor γt (RORyt); T Helper Cell (TH17)
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: 3+3 design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): XT-0528 250 mg administered once daily
  Interventions: Drug: XT-0528
- Cohort 2 (Experimental): XT-0528 500 mg administered once daily
  Interventions: Drug: XT-0528
- Cohort 3 (Experimental): XT-0528 1000 mg administered once daily
  Interventions: Drug: XT-0528
- Cohort 4 (Experimental): XT-0528 1500 mg administered once daily
  Interventions: Drug: XT-0528
- Cohort 5 (Experimental): XT-0528 2500 mg administered once daily
  Interventions: Drug: XT-0528

INTERVENTIONS:
Drug: XT-0528 — Once Daily

SUMMARY:
This study is an open-label, Phase 1, multicenter, continuous dose escalation study of XT-0528 in adult subjects with Advanced or Metastatic Solid Tumor Malignancies.

The study will consist of 4 periods:

Screening Period (up to 28 days prior to Cycle 1 Day 1) Safety Run-in Period (Cycle 1; continuous dosing on Days 1-21 of 28-day cycle) Continuous Dosing Period (Cycle 2 and beyond; continuous dosing on Days 1-28 of 28-day cycle) Safety Follow-up Period (30 days post-last dose).

DETAILED DESCRIPTION:
Primary Objective

* To determine the dose recommended for future Phase 2 studies (RP2D) that maximally suppresses T helper 17 (TH17) cell activities with an absence of dose limiting toxicity (DLT) and without exceeding the maximum tolerable dose (MTD).

Secondary Objective

* To establish the pharmacokinetics (PK) of orally administered XT-0528.
* To observe subjects for evidence of the antitumor activity of XT-0528.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 years of age at the time of consent;
2. Able to understand the key components of the study as described in the written informed consent document, and willing and able to provide written informed consent;
3. In the opinion of the Investigator, is able to adhere to the requirements of the study;
4. Willing and able to comply with the contraceptive requirements of the study:

   1. If female, is premenarcheal, surgically sterile (post hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), postmenopausal (>12 months of amenorrhea without alternative medical causes), or, if of childbearing potential, is using a highly effective method of contraception (combined estrogen/progestogen or progestogen-only hormonal contraceptives associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion/ligation, vasectomized partner[s], double barrier method [male condom with either cap, diaphragm or sponge with spermicide], or true abstinence of heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject [periodic abstinence , eg, calendar, ovulation, symptothermal, post-ovulation methods, and withdrawal, are not acceptable methods of contraception]), and agrees to continued use of this method until 120 days after the EOS Visit.
   2. If male, is vasectomized and has received medical assessment of surgical success, has undergone bilateral orchidectomy, or agrees to use an approved method of contraception (true abstinence of heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject, double barrier method [male condom with either cap, diaphragm or sponge with spermicide], female partner's use of a highly effective method of contraception, female partner is postmenopausal, or female partner is surgically sterile) and agrees to use this method until 120 days after the End of Study (EOS) Visit.
5. Subject must have histologically confirmed solid tumor malignancy that is metastatic or unresectable and have no additional approved standard of care treatment options, in the opinion of the Investigator;
6. Subject must have at least one biopsy accessible tumor;

   1. Subject must have at least one radiographically measurable lesion as per RECIST v1.1 defined as a lesion that is ≥10 mm in longest diameter or lymph node that is ≥15 mm in short axis as imaged by computed tomography (CT) scan or magnetic resonance imaging (MRI);
   2. Subject must be willing to undergo screening and on-study tumor biopsy. Note: if archival tissue from the identified tumor is available from a previous clinical biopsy (within the past year), a screening biopsy will not be required;
7. Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2;
8. Subject must have an anticipated life expectancy >3 months;
9. Subject must have normal organ and bone marrow function within 14 days of initiating study drug as defined below:

   1. Absolute neutrophil count ≥1,500/mcL;
   2. Platelets ≥100,000/mcL;
   3. Total bilirubin <1.5 × ULN (except known Gilbert's syndrome);
   4. Aspartate aminotransferase (AST) [serum glutamic-oxaloacetic transaminase SGOT)]/ Alanine aminotransferase (ALT) [serum glutamic-pyruvic transaminase (SGPT)] ≤2.5 × upper limit of normal (ULN);
   5. Creatinine clearance ≥60 mL/min/1.73 m2 calculated using the Cockcroft-Gault (C-G) equation.
10. Subjects must have resolution (Grade ≤1 or returned to baseline) of toxic effect(s) of the most recent prior therapy except:

    1. Grade 2 alopecia and Grade 2 fatigue, for which resolution is not required;
    2. Grade 2 elevation of AST, ALT or total bilirubin for patients with liver metastasis who started treatment with Grade 2 AST/ALT/total bilirubin and the highest increase was <50% relative to baseline and lasted for less than 1 week.
11. Subjects who received major surgery or radiation therapy of >30 Gy, must have recovered from the toxicity and/or complications from the intervention.

Exclusion Criteria:

1. Received other recent antitumor therapy including:

   1. Investigational therapy administered within the 28 days or 5 half-lives, whichever is shorter, prior to the first scheduled day of dosing in this study;
   2. Radiation or other standard systemic therapy within 14 days prior to the first scheduled dose in this study, including, in addition (if necessary), the timeframe for resolution of any actual or anticipated toxicities from such radiation.
2. Subject is expected to require any other form of antineoplastic therapy while on study;
3. Subject with active autoimmune disease requiring disease modifying therapy;
4. Subject has known history of prior malignancy except subjects who have undergone potentially curative therapy with no evidence of that disease recurrence within 5 years of therapy initiation. Allowable active malignancies include basal cell carcinoma, squamous cell (skin) carcinoma, or indolent lymphoma/leukemia not requiring treatment.
5. Subject requiring concurrent systemic corticosteroid therapy >10 mg/day of prednisone;
6. Subject with known active hepatitis B/C infection (positive viral titers) that has not been treated;
7. Subjects with known uncontrolled Human Immunodeficiency Virus (HIV)/Acquired Immunodeficiency Syndrome (AIDS) on anti-retroviral therapy defined by a cluster of differentiation 4 (CD4) count <200;
8. Subject has known central nervous system, meningeal, or epidural disease. Subjects with stable brain metastases for at least 4 weeks following definitive local treatment without new or enlarging brain metastases are eligible if corticosteroid requirement is ≤7.5 mg/day of prednisone (or equivalent);
9. Subject with a known history of significant cardiovascular disease as evidence by New York Heart Association (NYHA) classification Stage III/IV heart failure, unstable angina, myocardial infarction within the past 6 months, or uncontrolled arrhythmias;
10. Subjects has known history of corrected QT Interval (QTc) prolongation or observed QTc prolongation >470 ms during screening ECG;
11. Subject with known history of gastrointestinal (GI) disease that could affect drug absorption (eg, malabsorptive disorders, inflammatory bowel disease, short bowel from significant bowel resection, intestinal obstruction for peritoneal carcinomatosis);
12. Subject with known history or presence of allergic or adverse response to XT-0528 or related drugs or its excipients;
13. Subject requires use of strong inhibitors, strong inducers, and sensitive substrates of major cytochrome P450 enzymes (CYP) and drug transporters.
14. Subjects requiring chronic use of acid reducing agents (ARAs) are excluded from the study unless able to suspend use of ARAs for 48 hours prior to PK sampling days
15. Subject is pregnant, plans to become pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of study participation;
16. Subject has known psychiatric or substance abuse disorder(s) that would interfere with cooperation with required elements of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To determine the dose recommended for future Phase 2 studies (RP2D) that maximally suppresses Th17 cell activities | Cycle 1 (Days 1-21)
  Determination of Th17 cell suppression by measuring serum levels of Th17 cytokines before and during continuous dosing of XT-0528
To determine the dose recommended for future Phase 2 studies (RP2D) with an absence of dose limiting toxicity (DLT) and without exceeding the maximum tolerable dose (MTD). | Cycle 1 (Days 1-21)
  Determination of MTD, in the continuous dosing setting, as assessed by collection of adverse event/serious adverse event (AE/SAE) information, if MTD is reached during dose escalation.

SECONDARY OUTCOMES:
To establish the pharmacokinetics (PK) of orally administered XT-0528 and its (R)-isomer - Cmax | End of Cycle 1 (Days 1-21 of 28-day Cycle)
  maximum plasma concentration (Cmax)
To establish the pharmacokinetics (PK) of orally administered XT-0528 and its (R)-isomer - Cmax Steady State | End of Cycle 1 (Days 1-21 of 28-day Cycle)
  maximum plasma concentration at steady state (Cmax,ss)
To establish the pharmacokinetics (PK) of orally administered XT-0528 and its (R)-isomer - Tmax | End of Cycle 1 (Days 1-21 of 28-day Cycle)
  time to Cmax (Tmax)
To establish the pharmacokinetics (PK) of orally administered XT-0528 and its (R)-isomer - Tmax Steady State | End of Cycle 1 (Days 1-21 of 28-day Cycle)
  time to Cmax at Steady State (Tmax,ss)
To establish the pharmacokinetics (PK) of orally administered XT-0528 and its (R)-isomer - AUC | End of Cycle 1 (Days 1-21 of 28-day Cycle)
  area under the concentration-time curve calculated using linear trapezoidal rule from time zero to 24 hours, the dosing interval, after first dose (AUC0-t)
To establish the pharmacokinetics (PK) of orally administered XT-0528 and its (R)-isomer - AUC Steady State | End of Cycle 1 (Days 1-21 of 28-day Cycle)
  area under the concentration-time curve calculated using linear trapezoidal rule from time zero to 24 hours, the dosing interval, after first dose at Steady State (AUC0-tau)
To observe subjects for evidence of the antitumor activity of XT-0528 - ORR | End of Cycle 3 (Each cycle is 28 days)
  To determine the objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. * Overall response rate (ORR) is defined as the proportion of participants whose best observed response is either a complete response (CR) or partial response (PR) per RECIST in the population of interest
To observe subjects for evidence of the antitumor activity of XT-0528 - PFS | End of Cycle 3 (Each cycle is 28 days)
  To determine the median progression-free survival (PFS). Progression free survival (PFS) for a participant is defined as the time from first dosing date to the date of the first objectively documented disease progression per RECIST in the population of interest, or death due to any cause, whichever occurs first
To measure anti-drug antibody (ADA) formation against XT-0528 | End of Cycle 3 (Each cycle is 28 days)
  Neutralizing antibody assessments will be performed in samples positive for ADA and will be analyzed to determine impact on rate and severity treatment-emergent adverse event(s) (TEAE).
To observe subjects for evidence of the antitumor activity of XT-0528 - OS | End of Cycle 3 (Each cycle is 28 days)
  To determine the median overall survival (OS). Overall survival (OS) is defined as the time from enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Kelley, MD, Study Director — Xenthera, Inc.

IPD SHARING:
Plan to Share IPD: No
There are no plans to share information at this time.